CLINICAL TRIAL: NCT05513586
Title: A Phase 3, Open-label, Non-controlled, Extension Study to Evaluate the Long-term Safety of TAK-771 in Japanese Patients With Primary Immunodeficiency Disease (PID)
Brief Title: A Study to Evaluate the Long-term Safety of TAK-771 in Japanese Primary Immunodeficiency Disease (PID) Participants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-771-3005; jRCT2041220059 (Registry Identifier: jRCT)
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Primary Immunodeficiency Diseases (PID)
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAK-771 (Experimental): TAK-771 includes Immune Globulin Infusion (IGI) 10% and Recombinant Human Hyaluronidase (rHuPH20). Participants will receive SC infusion of rHuPH20 solution at a dose of 80 U/g IgG first, followed by SC infusion of 10% IGI within 10 minutes of completion of the infusion of rHuPH20 solution.
  Interventions: Drug: TAK-771

INTERVENTIONS:
Drug: TAK-771 — Immune Globulin Infusion (IGI) 10% and Recombinant Human Hyaluronidase (rHuPH20)
  Other Names: Immune Globulin Infusion 10% (Human) with Recombinant Human Hyaluronidase

SUMMARY:
The main aim of the study is to check side effect from the study treatment with TAK-771 in long term.

Participants can have taken part in the previous study TAK-771-3004 (NCT05150340). For those who can take part, the participants will receive injections of TAK-771 after the end of the previous study. The participants will be treated with TAK-771 for totally 3 years.

There will be many clinic visits. The number of visits will depend on the infusion cycles of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Participant have completed or is about to complete Study TAK-771-3004 (NCT05150340).
2. Written and/or electronic informed consent is obtained from either the participant or the participant's legally authorized representative prior to any study-related procedures and study product administration. If a participant is <18 years of age, written and/or electronic informed consent should also be obtained from the participant's legally authorized representative in addition to written informed assent by a participant if appropriate.
3. Participant is willing and able to comply with the requirements of the protocol.

Exclusion Criteria:

1. Participant has developed a new serious medical condition during Study TAK-771-3004 such that the participant's safety or medical care would be impacted by participation in the study.
2. Participant is willing to participate in other clinical trials.
3. Women of childbearing potential who meet any one of the following criteria:

   1. Participant presents with a positive pregnancy test.
   2. Participant does not agree to employ adequate birth-control measures (eg, intrauterine device, condom [for male partner], or birth-control pills) throughout the course of the study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Treatment-Emergent Adverse Events (TEAEs) | Up to 3 years
  TEAEs are defined as AEs with onset after date-time of first dose of investigational drug or medical conditions present prior to the start of investigational drug but increased in severity or relationship after date-time of first dose of investigational drug.
Percentage of Participants who Develop Anti-rHuPH20 Binding Antibody Titers of Greater Than or Equal to 1:160 and who Develop Neutralizing Antibodies to rHuPH20 | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (9):
- Japan (9):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Hospital of University of Occupational and Environmental Health, Kitakyushu, Fukuoka
  - Gifu University Hospital, Gifu, Gifu
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Kanagawa Children's Medical Center, Yokohama, Kanagawa
  - Saitama Prefectual Children's Medical Center, Saitama, Saitama
  - Shizuoka Childrens Hospital, Shizuoka, Shizuoka
  - Tokyo Medical Dental University Hospital, Bunkyo-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/972f9fef5a9d434a